CLINICAL TRIAL: NCT04041674
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of a Prime-boost Vaccine Regimen of GEO-D02 DNA and MVA/HIV62B With and Without B63521^11 gp120 and IHV01 gp120 Env Proteins in Healthy, HIV-uninfected Adult Participants *Imatinib Mesylate Per Oral as a Clinical Therapeutic for TB
Brief Title: Evaluating the Safety and Immunogenicity of a Prime-boost Vaccine Regimen of GEO-D02 DNA and MVA/HIV62B With and Without B63521^11 gp120 and IHV01 gp120 Env Proteins in Healthy, HIV-uninfected Adult Participants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Protocol undergoing additional revisions.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: HIV Vaccine Trials Network (HVTN), Fred Hutch / University of Washington (Unknown); GeoVax Labs, Inc (Unknown); Duke University (Other); University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HVTN 132; 34571 (Registry Identifier: DAIDS ES-Registry Number)
Record Dates: First submitted 2019-07-31; First posted 2019-08-01 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group 1 (T1): DNA + MVA + Placebo (IM) (Experimental): Participants will receive 3 mg of GEO-D02 DNA by intramuscular (IM) injection at Months 0 and 2.
  Participants will also receive 1×10^8 50% tissue culture infective dose (TCID50) of MVA/HIV62B plus placebo for B63521^11 gp120 plus placebo for IHV01, each by IM injection at Months 4, 6, and 10.
  Interventions: Biological: GEO-D02 DNA; Biological: MVA/HIV62B Vaccine; Biological: Protein Placebo
- Group 2 (T1): DNA + MVA + Placebo (SC) (Experimental): Participants will receive 3 mg of GEO-D02 DNA by IM injection at Months 0 and 2.
  Participants will also receive 1×10^8 TCID50 of MVA/HIV62B by IM injection plus placebo for B63521^11 gp120 by subcutaneous (SC) injection plus placebo for IHV01 by SC injection at Months 4, 6, and 10.
  Interventions: Biological: GEO-D02 DNA; Biological: MVA/HIV62B Vaccine; Biological: Protein Placebo
- Group 3 (T2): DNA + MVA + IHV01 + B63 (Experimental): Participants will receive 3 mg of GEO-D02 DNA by IM injection at Months 0 and 2.
  Participants will also receive 1×10^8 TCID50 of MVA/HIV62B plus 150 mcg of B63521^11 gp120 plus 150 mcg of IHV01, each by IM injection at Months 4, 6, and 10.
  Interventions: Biological: GEO-D02 DNA; Biological: MVA/HIV62B Vaccine; Biological: B63521^11 gp120; Biological: IHV01 Protein
- Group 4 (T3): DNA + MVA +IHV01 + Placebo (Experimental): Participants will receive 3 mg of GEO-D02 DNA by IM injection at Months 0 and 2.
  Participants will also receive 1×10^8 TCID50 of MVA/HIV62B plus placebo for B63521^11 gp120 plus 150 mcg of IHV01, each by IM injection at Months 4, 6, and 10.
  Interventions: Biological: GEO-D02 DNA; Biological: MVA/HIV62B Vaccine; Biological: IHV01 Protein; Biological: Protein Placebo
- Group 5 (T4): DNA + MVA +IHV01 (SC)+ B63 (SC) (Experimental): Participants will receive 3 mg of GEO-D02 DNA by IM injection at Months 0 and 3.
  Participants will also receive 1×10^8 TCID50 of MVA/HIV62B by IM injection plus 150 mcg of B63521^11 gp120 by SC injection plus 150 mcg of IHV01 by SC injection at Months 4, 6, and 10.
  Interventions: Biological: GEO-D02 DNA; Biological: MVA/HIV62B Vaccine; Biological: B63521^11 gp120; Biological: IHV01 Protein

INTERVENTIONS:
Biological: GEO-D02 DNA — Administered by IM injection into the vastus lateralis
Biological: MVA/HIV62B Vaccine — Administered by IM injection into the vastus lateralis
Biological: B63521^11 gp120 — Administered as a IM or SC injection into the vastus lateralis or overlying subcutaneous tissue as the MVA dose
  Arms: Group 3 (T2): DNA + MVA + IHV01 + B63; Group 5 (T4): DNA + MVA +IHV01 (SC)+ B63 (SC)
Biological: IHV01 Protein — Administered as a IM or SC injection into the vastus lateralis or overlying subcutaneous tissue as the MVA dose
  Arms: Group 3 (T2): DNA + MVA + IHV01 + B63; Group 4 (T3): DNA + MVA +IHV01 + Placebo; Group 5 (T4): DNA + MVA +IHV01 (SC)+ B63 (SC)
Biological: Protein Placebo — Sodium Chloride for Injection, 0.9% USP
  Administered as a IM or SC injection into the vastus lateralis or overlying subcutaneous tissue as the MVA dose
  Arms: Group 1 (T1): DNA + MVA + Placebo (IM); Group 2 (T1): DNA + MVA + Placebo (SC); Group 4 (T3): DNA + MVA +IHV01 + Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of a prime-boost vaccine regimen of GEO-D02 DNA and MVA/HIV62B with and without B63521^11 gp120 and IHV01 gp120 Env proteins in healthy, HIV-uninfected adult participants.

DETAILED DESCRIPTION:
This study will evaluate the safety and immunogenicity of a prime-boost vaccine regimen of GEO-D02 DNA and MVA/HIV62B with and without B63521^11 gp120 and IHV01 gp120 Env proteins in healthy, HIV-uninfected adult participants.

Participants will be randomly assigned to one of five groups. Participants in all five groups will receive GEO-D02 DNA by intramuscular (IM) injection at Months 0 and 2. Then, at Months 4, 6, and 10, participants will receive three additional injections according to their assigned group:

* Group 1: MVA/HIV62B, placebo for B63521^11 gp120, and placebo for IHV01, all by IM injection
* Group 2: MVA/HIV62B by IM injection and placebo for B63521^11 gp120 and for IHV01, both by subcutaneous (SC) injection
* Group 3: MVA/HIV62B, B63521^11 gp120, and IHV01, all by IM injection
* Group 4: MVA/HIV62B, placebo for B63521^11 gp120, and IHV01, all by IM injection
* Group 5: MVA/HIV62B by IM injection and IHV01 and B63521^11 gp120, both by SC injection

Participants will attend several study visits through Month 16. Visits may include physical examinations, blood and urine collection, electrocardiogram, HIV testing, risk reduction counseling, and questionnaires. Study staff will contact participants at Month 24 for follow-up health monitoring.

ELIGIBILITY:
Inclusion Criteria

General and Demographic Criteria

* Age of 18 to 50 years
* Access to a participating HVTN Clinical Research Site (CRS) and willingness to be followed for the planned duration of the study
* Ability and willingness to provide informed consent
* Assessment of understanding: volunteer demonstrates understanding of this study; completes a questionnaire prior to first vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Willing to be contacted after completion of scheduled clinic visits for a total of 2 years following initial study injection
* Agrees not to enroll in another study of an investigational research agent while in this study
* Good general health as shown by medical history, physical exam, and screening laboratory tests

HIV-Related Criteria:

* Willingness to receive HIV test results
* Willingness to discuss HIV infection risks and amenable to HIV risk reduction counseling
* Assessed by the clinic staff as being at "low risk" for HIV infection and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit (see the study protocol).

Laboratory Inclusion Values

Hemogram/Complete blood count (CBC)

* Hemoglobin greater than or equal to 11.0 g/dL for volunteers who were assigned female sex at birth, greater than or equal to 13.0 g/dL for volunteers who were assigned male sex at birth. For transgender participants who have been on hormone therapy for more than 6 consecutive months, determine hemoglobin eligibility based on the gender with which they identify (ie, a transgender female who has been on hormone therapy for more than 6 consecutive months should be assessed for eligibility using the hemoglobin parameters for persons assigned female sex at birth).
* White blood cell count equal to 2,500 to 12,000 cells/mm^3 with normal differential, or differential approved by Investigator of Record (IoR) as not clinically significant
* Total lymphocyte count greater than or equal to 650 cells/mm^3 with normal differential, or differential approved by IoR as not clinically significant
* Remaining differential either within institutional normal range or with site physician approval
* Platelets equal to 125,000 to 550,000 cells/mm^3

Chemistry

* Chemistry panel: alanine aminotransferase (ALT) less than 1.25 times the institutional upper limit of normal; creatinine less than or equal to 1.1 times the institutional upper limits of normal.

HIV Status

* Negative HIV-1 and -2 blood test: US volunteers must have a negative U.S. Food and Drug Administration (FDA)-approved enzyme immunoassay (EIA).

Urine

* Normal urine:

  * Negative or trace urine protein, and
  * Negative, trace, or 1+ blood urine hemoglobin (if +1 hemoglobin is present on dipstick, a microscopic urinalysis with red blood cells levels within institutional normal range).

Reproductive Status

* Volunteers who were assigned female sex at birth: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test at screening (ie, prior to randomization) and prior to study product administration on the day of study product administration. Persons who are NOT of reproductive potential due to having undergone hysterectomy or bilateral oophorectomy (verified by medical records), are not required to undergo pregnancy testing.
* Reproductive status: A volunteer who was assigned female sex at birth:

  * Must agree to consistently use effective contraception (see the study protocol) for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment until 3 months after the final study vaccination. Effective contraception is defined as using the following methods:

    * Condoms (male or female) with or without a spermicide,
    * Diaphragm or cervical cap with spermicide,
    * Intrauterine device (IUD),
    * Hormonal contraception,
    * Tubal ligation, or
    * Any other contraceptive method approved by the HVTN 132 Protocol Safety Review Team (PSRT)
    * Successful vasectomy in any partner assigned male sex at birth (considered successful if a volunteer reports that a male partner has [1] documentation of azoospermia by microscopy, or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity postvasectomy);
  * Or not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy, or bilateral oophorectomy;
  * Or be sexually abstinent.
* Volunteers who were assigned female sex at birth must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit.

Exclusion Criteria

* Blood products received within 120 days before first vaccination.
* Investigational research agents received within 30 days before first vaccination.
* Body mass index (BMI) greater than or equal to 40.
* Volunteer has 2 or more of the following cardiac risk factors:

  * Participant report of history of elevated blood cholesterol defined as fasting low-density lipoprotein (LDL) greater than 160 mg/dL;
  * First degree relative (eg, mother, father, brother, or sister) who had coronary artery disease before the age of 50 years;
  * Current smoker; or
  * BMI greater than or equal to 35.
* Intent to participate in another study of an investigational research agent or any other study that requires non-HVTN HIV antibody testing during the planned duration of the HVTN 132 study.
* Pregnant or breastfeeding.
* Active duty and reserve US military personnel.

Vaccines and other Injections

* Smallpox vaccine received within the last 5 years.
* HIV vaccine(s) received in a prior HIV vaccine trial. For volunteers who have received control/placebo in an HIV vaccine trial, the HVTN 132 PSRT will determine eligibility on a case-by-case basis.
* Non-HIV experimental vaccine(s) received within the last 1 year in a prior vaccine trial. Exceptions may be made by the HVTN 132 PSRT for vaccines that have subsequently undergone licensure by the FDA or by the national regulatory authority where the volunteer is enrolling. For volunteers who have received control/placebo in an experimental vaccine trial, the HVTN 132 PSRT will determine eligibility on a case-by-case basis. For volunteers who have received an experimental vaccine(s) greater than 1 year ago, eligibility for enrollment will be determined by the HVTN 132 PSRT on a case-by-case basis.
* Live attenuated vaccines received within 30 days before first study injection or scheduled within 14 days after the first study injection (eg, measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever; live attenuated influenza vaccine.)
* Any vaccines that are not live attenuated vaccines and were received within 14 days prior to first vaccination (eg, tetanus, pneumococcal, Hepatitis A or B.)
* Allergy treatment with antigen injections within 30 days before first vaccination or that are scheduled within 14 days after first vaccination.

Immune System

* Immunosuppressive medications received within 168 days before first vaccination (Not exclusionary: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatologic condition; or [4] a single course of oral/parenteral prednisone or equivalent at doses less than or equal to 60 mg/day and length of therapy less than 11 days with completion at least 30 days prior to enrollment.)
* Serious adverse reactions to vaccines or to vaccine components such as mannitol, aluminum hydroxide, and egg products, including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded from participation: a volunteer who had a non-anaphylactic adverse reaction to pertussis vaccine as a child.)
* Immunoglobulin received within 60 days before first vaccination.
* Autoimmune disease, current or history (Not exclusionary: mild, well-controlled psoriasis.)
* Immunodeficiency.

Cardiac

* History of myocarditis, pericarditis, cardiomyopathy, congestive heart failure with permanent sequelae, clinically significant arrhythmia (including any arrhythmia requiring medication, treatment, or clinical follow-up.)
* Electrocardiography (ECG) with clinically significant findings, or features that would interfere with the assessment of myo/pericarditis, as determined by a contract ECG Lab or cardiologist, including any of the following: (1) conduction disturbance (complete left or complete right bundle branch block or nonspecific intraventricular conduction disturbance with QRS greater than or equal to 120 ms, PR interval greater than or equal to 220ms, any second or third degree atrioventricular (AV) block, or QTc prolongation (greater than 450ms)); (2) repolarization (ST segment or T wave) abnormality that will interfere with the assessment of myo/pericarditis; (3) significant atrial or ventricular arrhythmia; (4) frequent atrial or ventricular ectopy (eg, frequent premature atrial contractions, 2 premature ventricular contractions in a row); (5) ST elevation consistent with ischemia; (6) evidence of past or evolving myocardial infarction.

Clinically significant medical conditions

* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

  * A process that would affect the immune response,
  * A process that would require medication that affects the immune response,
  * Any contraindication to repeated injections or blood draws,
  * A condition that requires active medical intervention or monitoring to avert grave danger to the volunteer's health or well-being during the study period,
  * A condition or process for which signs or symptoms could be confused with reactions to vaccine, or
  * Any condition specifically listed among the exclusion criteria below.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a volunteer's ability to give informed consent.
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
* Current anti-tuberculosis (TB) prophylaxis or therapy.
* Asthma other than mild or moderate, well-controlled asthma. (Symptoms of asthma severity as defined in the most recent National Asthma Education and Prevention Program (NAEPP) Expert Panel report.) Exclude a volunteer who:

  * Uses a short-acting rescue inhaler (typically a beta 2 agonist) daily, or
  * Uses high dose inhaled corticosteroids, or
  * In the past year has had either of the following:

    * Greater than 1 exacerbation of symptoms treated with oral/parenteral corticosteroids;
    * Needed emergency care, urgent care, hospitalization, or intubation for asthma.
* Diabetes mellitus type 1 or type 2 (Not exclusionary: type 2 cases controlled with diet alone or a history of isolated gestational diabetes.)
* Thyroidectomy, or thyroid disease requiring medication during the last 12 months. (Not exclusionary: well-controlled non-autoimmune thyroid disease.)
* Hypertension:

  * If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined in this protocol as consistently less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be less than or equal to 150 mm Hg systolic and less than or equal to 100 mm Hg diastolic. For these volunteers, blood pressure must be less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic at enrollment.
  * If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure greater than or equal to 150 mm Hg at enrollment or diastolic blood pressure greater than or equal to 100 mm Hg at enrollment.
* Bleeding disorder (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions.)
* Malignancy (Not excluded from participation: Volunteer who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure, or who is unlikely to experience recurrence of malignancy during the period of the study.)
* Seizure disorder: History of seizure(s) within past three years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
* Asplenia: any condition resulting in the absence of a functional spleen.
* History of generalized urticaria, angioedema, or anaphylaxis. (Not exclusionary: angioedema or anaphylaxis to a known trigger with at least 5 years since last reaction to demonstrate satisfactory avoidance of trigger.)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of local reactogenicity signs and symptoms | Measured through Month 10
  Local symptoms include pain and/or tenderness at the injection site.
Frequency of systemic reactogenicity signs and symptoms | Measured through Month 10
  Systemic symptoms include increased body temperature, malaise and/or fatigue, myalgia, headache, chills, arthralgia, and nausea.
Frequency of adverse events | Measured through Month 16
  Summarized using Medical Dictionary for Regulatory Activities (MedDRA) System Organ Class and preferred terms
Frequency of serious adverse events | Measured through Month 16
  Summarized using MedDRA System Organ Class and preferred terms
HIV-specific IgG binding magnitude to cross-clade panels of gp120 and V1V2, and gp41 | Measured through Month 10.5
  As assessed by binding antibody multiplex assay (BAMA)
HIV-specific IgG binding response rate to cross-clade panels of gp120 and V1V2, and gp41 | Measured through Month 10.5
  As assessed by BAMA
HIV-specific IgG binding breadth to cross-clade panels of gp120 and V1V2, and gp41 | Measured through Month 10.5
  As assessed by BAMA
Response rate of CD4+ T-cell responses to Env | Measured through Month 10.5
  As assessed by intracellular cytokine staining (ICS)
Magnitude of CD4+ T-cell responses to Env | Measured through Month 10.5
  As assessed by ICS

SECONDARY OUTCOMES:
HIV-specific IgG binding magnitude to V3, CD4i and gp41 IDR | Measured through Month 10.5
  As assessed by BAMA
HIV-specific IgG binding response rate to V3, CD4i and gp41 IDR | Measured through Month 10.5
  As assessed by BAMA
IgA responses to gp120, V1V2, and gp41 | Measured through Month 10.5
  As assessed by BAMA
IgG3 responses to gp120, V1V2, and gp41 | Measured through Month 10.5
  As assessed by BAMA
IgG avidity to defined epitope specificities | Measured through Month 10.5
  Determined from the immunogenicity data
HIV-specific IgG binding magnitude to gp120, V1V2, and gp41 | Measured through Month 16
  As assessed by BAMA
HIV-specific IgG binding response rate to gp120, V1V2, and gp41 | Measured through Month 16
  As assessed by BAMA
IgA responses to gp120 and gp41 | Measured through Month 16
  As assessed by BAMA
IgG3 responses to gp120 and gp41 | Measured through Month 16
  As assessed by BAMA
Response rate of antibody-dependent cellular cytotoxicity (ADCC)-mediating antibody responses | Measured through Month 16
  Assessed using serum samples taken at a primary immunogenicity timepoint
Magnitude of ADCC-mediating antibody responses | Measured through Month 16
  Assessed using serum samples taken at a primary immunogenicity timepoint
Response rate of antibody-dependent cellular phagocytosis (ADCP)-mediating antibody responses | Measured through Month 16
  Measured using serum samples taken at baseline and at a primary immunogenicity timepoint
Magnitude of antibody-dependent cellular phagocytosis (ADCP)-mediating antibody responses | Measured through Month 16
  Measured using serum samples taken at baseline and at a primary immunogenicity timepoint
Response rate of vaccine-elicited antibody binding to FcƴR proteins | Measured through Month 16
  Assessed on serum samples taken at the primary immunogenicity timepoints and baseline
Magnitude of vaccine-elicited antibody binding to FcƴR proteins | Measured through Month 16
  Assessed on serum samples taken at the primary immunogenicity timepoints and baseline

CONTACTS AND LOCATIONS:
Overall Officials: Michael Keefer, Study Chair — University of Rochester; Mark Pilkinton, Study Chair — Vanderbilt University

IPD SHARING:
Plan to Share IPD: No